CLINICAL TRIAL: NCT06213532
Title: CONNECTing to LungCare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other); Alere San Diego (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 226311; NCI-2023-10506 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Smoking Cessation; Cigarette Smoking-Related Carcinoma; Lung Carcinoma
MeSH Terms: conditions — Smoking Cessation; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: The first cohort of participants will be enrolled on the Beta Arm or intervention development. Once developed, new participants will be randomized into Groups 1 and Groups 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Beta testing (CONNECTing to LungCare, feedback) (Other): Participants interact with the CONNECTing to LungCare intervention and provide feedback in support of intervention refinement.
  Interventions: Behavioral: Smoking Cessation Intervention; Other: Survey Administration
- Feasibility trial, Group I (CONNECTing to LungCare) (Experimental): Participants receive the CONNECTing to LungCare intervention, including education about the benefits and risks of LCS and the importance of shared decision making, computerized assessments of the participant's smoking status, readiness to quit and concerns about quitting, and video segments tailored to the participant's responses to assessment questions, prior to their primary care appointment. Participants and their providers receive a tailored summary of the participant's concerns and barriers to quitting to enhance motivation for smoking cessation and shared decision-making discussions. Participants then receive up to 3 follow-up phone calls over 10-15 minutes each encouraging them to follow up with their provider, to complete the shared decision-making conversation, obtain LCS if appropriate, and access smoking cessation resources. Participants may also receive brief, tailored follow-up text messages that include links to video segments or cessation resources 1-3 times weekly.
  Interventions: Behavioral: Smoking Cessation Intervention; Other: Saliva Collection; Other: Survey Administration
- Feasibility trial, Group II (usual care) (Active Comparator): Participants receive usual care from their provider at their primary care appointment.
  Interventions: Behavioral: Smoking Cessation Intervention; Other: Saliva Collection; Other: Survey Administration

INTERVENTIONS:
Behavioral: Smoking Cessation Intervention — Multimedia program administered either remotely or in person
  Other Names: CONNECTing to LungCare intervention
Other: Saliva Collection — Saliva samples will be collected from each participant
  Other Names: Biospecimen Collection; Specimen Sample; Saliva Sample
  Arms: Feasibility trial, Group I (CONNECTing to LungCare); Feasibility trial, Group II (usual care)
Other: Survey Administration — Ancillary studies

SUMMARY:
This study evaluates a smoking cessation intervention (CONNECTing to LungCare) for improving shared decision-making conversations about smoking cessation and lung cancer screening between patients and providers. Shared decision making is a patient care model in which providers offer information regarding risks and benefits, patients express their values and preferences, and then healthcare decisions are jointly discussed between the patient and provider. Patient education, aided by decision support tools, can increase patients' knowledge, decrease their decisional conflict, promote decision making, and improve the patients' perception of risk. CONNECTing to LungCare is an interactive education intervention that addresses lung cancer screening and smoking cessation and provides participants with a tailored summary that may make them more likely to have shared decision-making discussions with their providers about smoking cessation and lung cancer screening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Aim 1: Development of the smoking cessation and LCS intervention, CONNECTing to LungCare.

Aim 2: Test CONNECTing to Lung Care for Feasibility and Acceptability (N=120)

Aim 3: To qualitatively evaluate feasibility and acceptability of the intervention and study procedures from the perspectives of patients, providers, staff and administrators and other stakeholders.

OUTLINE:

BETA TESTING: Participants interact with the CONNECTing to LungCare intervention and provide feedback in support of intervention refinement.

FEASIBILITY TRIAL: Participants are randomized to 1 of 2 groups.

GROUP I: Participants receive the CONNECTing to LungCare intervention, including education about the benefits and risks of LCS and the importance of shared decision making, computerized assessments of the participant's smoking status, readiness to quit and concerns about quitting, and video segments tailored to the participant's responses to assessment questions, prior to their primary care appointment. Participants and their providers receive a tailored summary of the participant's concerns and barriers to quitting to enhance motivation for smoking cessation and shared decision making discussions. Participants then receive up to 3 follow-up phone calls over 10-15 minutes each encouraging them to follow up with their provider, to complete the shared decision-making conversation, obtain LCS if appropriate, and access smoking cessation resources. Participants may also receive brief, tailored follow-up text messages that include links to video segments or cessation resources 1-3 times weekly.

GROUP II: Participants receive usual care from their provider at their primary care appointment.

After completion of study intervention, participants are followed up at 1 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* English, Spanish and Cantonese speaking
* Age >= 18 years old
* Primary care patients at the University of California, San Francisco (UCSF) General Internal Medicine (GIM) clinics
* Must be current smokers and/or candidates for Lung Cancer Screening (LCS).

Key Informant Interviews:

- Must be working in one of the clinics participating in CONNECTing to LungCare.

Exclusion Criteria:

* Not a current smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Up to 1 year
  The percentage of participants who were contacted and joined the study will be reported.
Retention rates | Up to 1 year
  The percentage of participants who joined the study and completed the program will be reported.
Adherence rates | Up to 1 year
  The percentage of participants who joined the study and completed all tasks within the program will be reported.
Overall time required to recruit to the target sample size (Feasibility Cohort) | Up to 1 year
  The overall time in weeks required to recruit participants for the feasibility cohort will be reported.
Number of eligible participants | Up to 1 year
  The number of eligible participants required to recruit the required sample size will be reported

SECONDARY OUTCOMES:
Smoking cessation rates | At 3 months
  Will evaluate the impact of the intervention on smoking cessation rates. Rates of smoking cessation will be measured by self-report and validated by salivary cotinine levels.
Lung cancer screening (LCS) rates | Up to 3 months
  Rates of LCS will be evaluated through review of the electronic health record (EHR)
Shared decision making about LCS | Up to 3 months
  Evidence of shared decision-making conversation will be obtained through one week follow up phone call and with review of the EHR three months after the primary care physician visit.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Walsh-Cassidy, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No